CLINICAL TRIAL: NCT03091881
Title: Attenuation of Spinal Induced Hypotension With Granisetron in Type I Diabetic Parturients
Brief Title: Granisetron in Diabetic Parturients Decrease Spinal Induced Hypotension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Mohamed A Elsadany, MD, Lecturer of anesthesiology, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2978
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Spinal-induced Hypotension
Keywords: Granisetron; Spinal induced hypotension
MeSH Terms: interventions — Granisetron

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Granisetron group (Active Comparator): patients in this group will receive intravenous Granisetron 0.1 MG/ML 10 minutes before spinal anesthesia
  Interventions: Drug: Granisetron 0.1 MG/ML
- Placebo group (Placebo Comparator): Patients in this group will receive 10 ml normal saline as placebos considering the same timing and color of solution
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Granisetron 0.1 MG/ML — Granisetron 0.1 MG/ML Will be given 10 min before spinal block
  Other Names: Granisetron
  Arms: Granisetron group
Drug: Placebos — Placebos will be given 10 min before spinal block
  Other Names: Placebo
  Arms: Placebo group

SUMMARY:
Diabetic Parturients are exposed to intraoperative hypotension after spinal anesthesia and we proposed that intravenous Granisterone 1 mg will attenuate the hypotension occurred with spinal block during Cesarean sections.

DETAILED DESCRIPTION:
Introduction:

Spinal anesthesia is considered the first choice for cesarean sections if there are no absolute or relative contraindications. It is easy and has lower risks for mother and baby for most of cases. Anesthetists, especially junior staff, prefer spinal anesthesia for cesarean sections avoiding managing airway or inserting an endotracheal tube which is usually difficult in full term pregnant woman.

Hypotension that follows spinal anesthesia usually occur due to blockade of sympathetic vasomotor activity that is accentuated by compression of the aorta and inferior vena cava by the gravid uterus when the patient is in the supine position.

It starts very soon after intrathecal injection of the local anesthetic and may extend till the end of the block putting the anesthesia team in an explanatory situation. The pathophysiology of spinal hypotension is mainly due to the sympathetic blockade predominating pararsympathetic power to dilating blood vessels and subsequent blood pooling in the dilated blood vessels (mainly venous side).

Sudden bradycardia can occur from shift in cardiac autonomic balance toward the parasympathetic system from activation of left ventricular mechanoreceptors or chemoreceptors Bezold Jarisch reflex (BJR) or from an increase in baroreflex activity.[1] Serotonin released during low-volume states has been suggested as a possible trigger for the BJR.[2] Granisetron is a 5-Hydoxy Tryptamine 3 (5-HT3) receptor antagonist that is very effective in preventing nausea and vomiting.

Diabetes mellitus is a widespread disease that increases the risk of cardiovascular diseases and intraoperative mortalities. Diabetes is associated with increased risk of perioperative hypotension due to autonomic neuron system dysfunction associated with micro and macro complications of long standing hyperglycemia. The effect of preganglionic sympathetic fibers and cardiac sympathetic innervation blockade occurring during spinal anesthesia on cardiac autonomic neurons function are expected to be different in diabetic patients from that of normal patients.

In a large cohort of patients with type 1 and type 2 diabetes, Ziegler et al. [3], using predefined heart rate variability (HRV) tests and spectral analysis of the R-R intervals, found that 25.3% of patients with type 1 diabetes and 34.3% of patients with type 2 diabetes had abnormal findings. Clinical symptoms of autonomic dysfunction may not appear until long after diabetes onset.

However, subclinical cardiac neuropathic dysfunction, manifested as changes in HRV, may be detected within 1 year of diagnosis in type II diabetes and within 2 years of diagnosis in type I diabetes .[4]

The incidence of hypotension defined as systolic blood pressure less than 90 mm Hg and bradycardia defined as heart rate less than 50 beat/minute are haemodynamic adverse effects of spinal anesthesia in non-obstetric patients has been reported to be 33% and 13% respectively.[5,6]

Aim of the work:

This study will investigate the effect of the antiemetic drug Granisetron (G Setron 1 mg in 1 ml ampule) in reducing the incidence of hypotension occurred with spinal anesthesia in type I diabetic patients arranged for cesarean sections.

Material and Methods:

This study will be randomized double blind where the anesthetists', data collectors and patients will be blinded to the assigned groups.

After hospital ethics committee approval and written informed consents, 68 type I diabetic patients scheduled for cesarean sections will participate in this study at Operation Theater of Suez Canal University Hospitals. All participating patients will be randomly classified into two equal groups, the (G) Granisetron group and the (P) Placebo group.

The primary outcome will be the incidence of Hypotension defined as SBP < 90 mmHg occurred with spinal anesthesia in type I diabetic patients arranged for caesarean sections.

A total of 68 type I diabetic full term pregnant women enrolled for caesarean section deliveries under spinal anesthesia will be included in this study. Approval of our institutional medical committee and a written consent from patients will be obtained. Inclusion criteria will include diabetic (Type I) ladies aged above 21 years old arranged for elective caesarean section under spinal anesthesia. Exclusion criteria will include any contraindications for spinal anesthesia (like bleeding diathesis or regional infection at site of neuroaxial block), known allergy to Granisetron or local anaesthetic (heavy bupivacaine, Marcaine Spinal 0.5% Heavy, 5mg/ml, AstraZeneca ampule), chronic hypertension, pregnancy induced hypertension, or congenital or rheumatic heart diseases, antepartum haemorrhage, Fetal destress or gestational age < 36 week.

All patients will be randomly classified in to two equal groups (34 patients in each): G group will receive 1 mg Granisetron (G Setron, 1 mg/ml Egyptian Pharmaceutical Company) intravenously diluted in 10 ml normal saline 10 minutes before spinal anesthesia, and P group will receive 10 ml normal saline N.S as placebo considering the same timing and color of solution. Randomization will be performed using a computer based random number generator and sealed envelopes will not be opened till an informed consent is obtained. The study will be double-blind as the anesthetists, data collectors and patients will not know the assignment groups. The syringes of Granisetron and placebo will be prepared by an anesthetist who will not be informed about the study protocol.

All patients will be infused with 500 ml lactated ringer intravenously IV. Premedication with 30 ml of a 0.15 molar solution of sodium citrate will be given orally 15-30 minutes before surgery in addition to Ranitidine ampule (Zantac) 50 mg diluted in 10 ml N.S given intravenously slowly. Base line heart rate (HR) and mean arterial blood pressure (MABP) readings will be measured just before spinal anesthesia. Spinal anesthesia will be performed in the sitting position using 25-gauge spinal needle (B BRAUN Co.) in L3-L4 or L4-L5 lumbar interspaces, 12.5 mg (2.5 ml volume) 0.5% hyperbaric Bupivcaine (Marcaine Spinal 0.5% Heavy, 5mg/ml, AstraZeneca ampule) will be injected intrathecally over 1 minute. After spinal anesthesia, parturient will be placed on the operating table in the supine position with 15° of left lateral tilt with supplemental oxygen through a face mask at 5 L per min.

Sensory level will be evaluated by testing for cold sensation, and motor block will be assessed according to Bromage scale after 5 min. HR and mean arterial blood pressure will be recorded every 3 min until the end of surgery.

Blood pressure will be measured every 3 min Ephedrine 10 mg boluses will be used until hypotension (Mean blood pressure above 65 mmHg) is controlled and then the predetermined protocol will be followed.

Maintenance fluid of lactated Ringer's solution will be given at a rate of 10 ml/kg/h in both groups during the surgical procedure. An additional rapid bolus infusion (100 ml) of lactated Ringer's will be pushed at each episode of hypotension. 10 mg ephedrine will be administered if MBP is less than 65 mmHg. A second dose of 10 mg ephedrine will be repeated if hypotension persisted 5 min or recurred. Phenylephrine will be considered if persistent hypotension not responding to ephedrine. If bradycardia occurred defined as HR lower than 60 beat per min 0.5 mg atropine will be considered unless it is associated with hypotension, if that ephedrine will be the choice.

Demographic data of all patients (Age, Height, Weight, BMI, duration of procedure, duration of diabetes, Glycosylated Hemoglubin, and parity) will be recorded. Incidence of hypotension will be calculated and compared in both groups. Other useful information as incidence of bradycardia (HR< 50 beat/minute) and atropine, ephedrine, and phenylephrine administered doses will be recorded.

Nausea and vomiting will be recorded using Verbal Descriptive Scale (VDS) [0 = no nausea, 1 = mild nausea, 2 = moderate nausea, 3 = frequent vomiting and 4 = severe vomiting] [7]

References

1. Butterworth J. Physiology of spinal anesthesia: What are the implications for management? Reg Anesth Pain Med 1998;23: 370-3.
2. Adams VR, Valley AW. Granisetron: The second serotonin-receptor antagonist. Ann Pharmacother 1995;29:1240-51.
3. Ziegler D, Dannehl K, Mühlen H, Spüler M, Gries FA. Prevalence of cardiovascular autonomic dysfunction assessed by spectral analysis, vector analysis, and standard tests of heart rate variation and blood pressure responses at various stages of diabetic neuropathy. Diabet Med 1992; 9: 806- 814 [PubMed]
4. Pfeifer MA, Weinberg CR, Cook DL, Reenan A, Halter JB, Ensinck JW, Porte D., Jr Autonomic neural dysfunction in recently diagnosed diabetic subjects Diabetes Care 1984; 7: 447- 453 [PubMed]
5. Carpenter RL, Caplan RA, Brown DL, Stephenson C, Wu R (1992) Incidence and risk factors for side effects of spinal anesthesia.Anesthesiology 76: 906-916.
6. Arndt JO, Bömer W, Krauth J, Marquardt B (1998) Incidence and time course of cardiovascular side effects during spinal anesthesia after prophylactic administration of intravenous fluids or vasoconstrictors.Anesth Analg 87: 347-354.
7. Rhodes VA, Watson PM, Johnson MH. Development of reliable and valid measures of nausea and vomiting. Cancer Nurs.1984;7:33-41

ELIGIBILITY:
Inclusion Criteria:

* Type I diabetic patients
* Parturients presented for Cesarean section

Exclusion Criteria:

* Contraindications for spinal anesthesia (like bleeding diathesis or regional infection at site of neuroaxial block)
* Known allergy to Granisetron or local anaesthetic (heavy bupivacaine, Marcaine Spinal 0.5% Heavy, 5mg/ml, AstraZeneca ampule)
* Pregnancy induced hypertension
* Congenital or rheumatic heart diseases
* Antepartum haemorrhage
* Fetal destress or gestational age < 36 week

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Total Ephedrine consumption | 60 minutes after spinal anesthesia
  Total Ephedrine consumption in mg

SECONDARY OUTCOMES:
Incidence of bradycardia | 60 minutes after spinal anesthesia
  Incidence of bradycardia with Heart Rate less than 50 beats / minutes
Incidence of hypotension | 60 minutes after spinal anesthesia
  incidence of hypotension with systolic blood pressure less than 90 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Elsadany, M.D, Study Director — Suez Canal University, Faculty of Medicine, Anesthesia and Intensive Care Department; Amr M Helmy, M.D, Study Director — Suez Canal University, Faculty of Medicine, Anesthesia and Intensive Care Department; Emad E Ahmed, M.D, Principal Investigator — Suez Canal University, Faculty of Medicine, Anesthesia and Intensive Care Department; Abdelrhman Alshawadfy, M.D, Principal Investigator — Suez Canal University, Faculty of Medicine, Anesthesia and Intensive Care Department
Locations (1):
- Suez Canal University, Faculty of Medicine, Anesthesia and Intensive Care Department, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Butterworth J. Physiology of spinal anesthesia: what are the implications for management? Reg Anesth Pain Med. 1998 Jul-Aug;23(4):370-3; discussion 384-7. doi: 10.1016/s1098-7339(98)90008-6. No abstract available. PMID 9690588
- [Background] Adams VR, Valley AW. Granisetron: the second serotonin-receptor antagonist. Ann Pharmacother. 1995 Dec;29(12):1240-51. doi: 10.1177/106002809502901211. PMID 8672830
- [Background] Ziegler D, Dannehl K, Muhlen H, Spuler M, Gries FA. Prevalence of cardiovascular autonomic dysfunction assessed by spectral analysis, vector analysis, and standard tests of heart rate variation and blood pressure responses at various stages of diabetic neuropathy. Diabet Med. 1992 Nov;9(9):806-14. doi: 10.1111/j.1464-5491.1992.tb01898.x. PMID 1473320
- [Background] Pfeifer MA, Weinberg CR, Cook DL, Reenan A, Halter JB, Ensinck JW, Porte D Jr. Autonomic neural dysfunction in recently diagnosed diabetic subjects. Diabetes Care. 1984 Sep-Oct;7(5):447-53. doi: 10.2337/diacare.7.5.447. PMID 6499637
- [Background] Carpenter RL, Caplan RA, Brown DL, Stephenson C, Wu R. Incidence and risk factors for side effects of spinal anesthesia. Anesthesiology. 1992 Jun;76(6):906-16. doi: 10.1097/00000542-199206000-00006. PMID 1599111
- [Background] Arndt JO, Bomer W, Krauth J, Marquardt B. Incidence and time course of cardiovascular side effects during spinal anesthesia after prophylactic administration of intravenous fluids or vasoconstrictors. Anesth Analg. 1998 Aug;87(2):347-54. doi: 10.1097/00000539-199808000-00021. PMID 9706929
- [Background] Rhodes VA, Watson PM, Johnson MH. Development of reliable and valid measures of nausea and vomiting. Cancer Nurs. 1984 Feb;7(1):33-41. No abstract available. PMID 6559094